CLINICAL TRIAL: NCT02061566
Title: National Taiwan University Hospital Yu-Lin Branch
Brief Title: Indoxyl Sulfate Induces Leukocyte-endothelial Interactions Through Up-regulation of ICAM-1 in Acute Kidney Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201310062RINA
Record Dates: First submitted 2014-02-11; First posted 2014-02-13 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Renal Function Disorder
Keywords: Acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum BUN, Cre, ICAM-1
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acute kidney injury: Acute kidney injury in ICU
- Non acute kidney injury: Non acute kidney injury

SUMMARY:
Indoxyl sulfate (IS) is an anionic uremic toxin that is accumulated in the serum of patients with uremia. In previous study, the investigators successfully induced AKI animal model. IS enhanced intercellular adhesion molecule-1 (ICAM-1) expression in IL-1β-treated human umbilical vein endothelial cells (HUVECs) that this may play a critical role in the progression of AKI. However, the molecular mechanisms of ICAM-1 expression in IS-treated IL-1β-treated HUVECs need to be elucidated. HUVECs incubated with 0.2 or 1 mM IS for 24 h did not cause cytotoxicity. The IL-1β-induced ICAM-1 expression in HUVECs was significantly enhanced by IS pretreatment. Furthermore, the regulation of adhesion molecule expression involves a complex array of intracellular signaling pathways including mitogen-activated protein kinase (MAPKs), reactive oxygen species (ROS) and transcriptional factors. A better understanding of this might provide important insights into the prevention of AKI.

DETAILED DESCRIPTION:
Over the past decade, acute kidney injury (AKI) has acquired much attention because of their potentially devastating problems in clinical medicine. When kidneys lost their filtering function, a lot of dangerous metabolites were accumulated in the body, including urea, nitrogenous waste products and uremic toxins. Indoxyl sulfate (IS) is an anionic uremic toxin that is accumulated in the serum of patients with uremia. In previous study, the investigators successfully induced AKI animal model. IS enhanced intercellular adhesion molecule-1 (ICAM-1) expression in IL-1β-treated human umbilical vein endothelial cells (HUVECs) that this may play a critical role in the progression of AKI. However, the molecular mechanisms of ICAM-1 expression in IS-treated IL-1β-treated HUVECs need to be elucidated. HUVECs incubated with 0.2 or 1 mM IS for 24 h did not cause cytotoxicity. The IL-1β-induced ICAM-1 expression in HUVECs was significantly enhanced by IS pretreatment. Furthermore, the regulation of adhesion molecule expression involves a complex array of intracellular signaling pathways including mitogen-activated protein kinase (MAPKs), reactive oxygen species (ROS) and transcriptional factors. A better understanding of this might provide important insights into the prevention of AKI.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients

Exclusion Criteria:

* Less than 20 years old

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AKI in ICU
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Renal function recovery (BUN, Cre) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsiang Chou, MD, Principal Investigator — NTUH Yun-Lin branch
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan